CLINICAL TRIAL: NCT06571357
Title: The Effect of Pranic Healing Based on Rogers' Therapeutic Touch Nursing Theory on Cardiorespiratory Indices and Pain Related to Venipuncture in Children
Brief Title: Effect of Pranic Healing on Cardiorespiratory Indices and Pain During Venipuncture in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Pouran Varvani Farahani, PhD student in Pediatric Nursing, Near East University , Faculty of Nursing, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PVF2024CAM001
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pain, Acute; Therapeutic Touch
Keywords: Phlebotomy; Pain Management; Therapeutic Touch; Nursing Theory
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants in this clinical trial will be randomly assigned to one of two groups: an experimental group receiving Pranic Healing and a control group receiving standard care. Both groups will be observed in parallel for the duration of the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: To minimize biased information, we employed a double-blind approach. The data will be collected by the researcher, and the statistician will be unaware of the groups; data will be analysed as variables x1 and x2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pranic Healing Intervention (Experimental): Participants in this group will receive the Pranic Healing intervention, based on Martha Rogers' Science of Unitary Human Beings, specifically focusing on the concept of "Nursing as Facilitation of Healing." The Pranic Healing intervention will follow the advanced protocol as conceptualized by Master Choa Kok Sui, including the following seven techniques:
  Sensitizing the hands Scanning the Aura Cleansing the Aura Increasing the receptivity Energizing with prana Stabilizing the projected prana Releasing
  The intervention will be applied in three stages: 5 minutes before, during, and 5 minutes after venipuncture.
  Interventions: Behavioral: Pranic Healing
- routine care (No Intervention): Participants in this group will receive routine care without any Pranic Healing intervention.

INTERVENTIONS:
Behavioral: Pranic Healing — The Pranic Healing intervention will be applied according to the advanced protocol by Master Choa Kok Sui, involving seven key techniques: sensitizing the hands, scanning the aura, cleansing the aura, increasing receptivity, energizing with prana, stabilizing the projected prana, and releasing. The intervention will take place in three stages: 5 minutes before, during, and 5 minutes after venipuncture.
  Other Names: Touch therapy
  Arms: Pranic Healing Intervention

SUMMARY:
The goal of this clinical trial is to evaluate whether Pranic healing, based on Rogers' therapeutic touch nursing theory, can reduce pain and improve cardiorespiratory indices during venipuncture in children. The main questions it aims to answer are:

Does Pranic healing reduce the pain experienced by children during venipuncture? How does Pranic healing affect cardiorespiratory indices, such as heart rate, respiratory rate, and arterial oxygen saturation, during and after venipuncture?

Researchers will compare the effects of Pranic healing to routine care (without Pranic healing) to determine its effectiveness.

Participants will:

Receive Pranic healing or routine care before, during, and after venipuncture Have their pain levels, heart rate, respiratory rate, and arterial oxygen saturation measured Be randomly assigned to either the intervention group (Pranic healing) or the control group (routine care) Have their pain and physiological responses monitored and recorded during the procedure

DETAILED DESCRIPTION:
Study Title: The Effect of Pranic Healing Based on Rogers' Therapeutic Touch Nursing Theory on Cardiorespiratory Indices and Pain Related to Venipuncture in Children: A Double-Blind Randomized Clinical Trial Study Purpose:This study will investigate the efficacy of Pranic healing, informed by Rogers' therapeutic touch nursing theory, in mitigating pain and enhancing cardiorespiratory indices in children undergoing venipuncture. The double-blind, randomized clinical trial will be conducted in the pediatric ward of Near East University Hospital, Northern Cyprus.

Study Subjects: Sample Size: 46 school-aged children, aged 6 to 12 years. Sampling Method:Convenience sampling followed by random block sampling. Groups: Experimental group (Pranic healing) and control group.

Sample size determination:

The statistical population of this research includes school-aged children admitted to one hospital in Northern Cyprus.

After obtaining consent, the children were randomly will be divided into the experimental and control groups. Then, a control and experimental group of 23 people will be formed by random block sampling method. In this method, blocks are formed based on the variables in question, and half of the intervention people and half of the control people are included in each block, the main goal in this method is to balance the number of participants in each of the groups. The four block randomization method will be used and the patients will be placed in experimental group groups (A) and control group (B), so that first 12 blocks of four and one block of two were prepared as follows: AABB, ABAB , ABBA, BBAA, BABA, BAAB, ABAB, AABB, BBAA, BAAB, BABA, ABBA, AB And then people will be assigned to two groups based on the list prepared in terms of A and B; This work is continuously repeated until the sample size is completed.

The samples of this research according to the sample size formula considering the 20% drop, there are 23 school-age children in each group. That have criteria for entering the research. The samples are divided into control and intervention groups using convenience sampling method. To minimize biased information, we employed a double-blind approach. The data will be collected by the researcher, and the statistician will be unaware of the groups; data will be analysed as variables x1 and x2.

Based on the study (Dehghani et al., 2019) and the mean comparison formula, the first type error level is 0.05, the power of the test is 80%, the sample size in each group is 19 people, which is 23 people in each group considering 20% dropout.

Tools of data collection:

To address the goals of the research, the data will be collected using questionnaires, Pain intensity scale, flow sheet, the intensive care monitor and a pulse oximeter.

A) The questionnaire for collecting demographic data on children and parents will be one of the tools utilized.

B) Pain intensity scale: The instrument used to measure pain will be Wong and Baker Facial Pain Scale. This scale is used in children aged 3 and older to rate pain severity (Yıldırım & Gerçeker, 2023). The child was asked to choose the face expressing their pain. It was presented in 1988 and 1996 by Wong and Baker and consists of six cartoon figures with experiences of no pain to the most severe pain that is crying. (0 to 5 or 0 to 10) (Hockenberry, 2019b) In this research, Wong and Baker Facial Pain Scale will be used in Turkish. )Appendix 2 (Wong and Baker Facial Pain Scale has been widely used and its validity and reliability have been proven in acute pain (Kamki et al., 2022) . Seval conducted a project to validate the Turkish version this tool in 2020, obtaining the internal consistency coefficient was 0.851 and the correlations was r =0.79 (Seval, 2020).

C) Children's pain assessment and measurement of cardiorespiratory indices, recording flow sheet: It consists of seven items. These questionnaires will be completed through observation by researcher in both groups.

D) The respiration rate of the child, pulse rate and arterial oxygen saturation will be measured using a pulse oximeter and intensive care monitor. Pulse oximetry will be valid, and to ensure the reliability of research tool, only one pediatric pulse oximeter will be used for all participants. Equivalent reliability method will be also used to evaluate the reliability of the monitor; its accuracy will be compared with another device each time before the intervention.

Intervention: Experimental Group: Pranic healing will be administered 5 minutes before, during, and 5 minutes after venipuncture. Control Group: Will receive routine care without additional intervention.

Implementation phase:

The present study is a clinical trial study. The research population is all children aged 6 to 12 admitted with a diagnosis in the children's department of Near East Hospital in Northern Cyprus. 46 samples of eligible children whose mothers are willing to participate in the study will be selected. The samples will be divided into two equal groups by random and Convenience sampling method. After explaining the purpose and how to do the work, written informed consent will be obtained from the mothers. The samples will be divided into Pranic healing therapy and control groups.

Demographic information questionnaire will be completed for each child. To perform the intervention, Pranic healing will be performed 5 minutes before and during the venipuncture and 5 minutes after in the experimental group. The researcher who will perform Pranic therapy is trained by a Pranic therapist. She has a certificate from World Pranic Healing Foundation (Appendix 4. ( In this study interventions, the intervention will be conducted in the privacy of the participant's room. The participants will be guided. They will lie on their backs on their hospital beds for the treatment. Prior to the treatment, they will be instructed to relax as fully as possible and a brief explanation of Pranic healing procedures will be given by an informative brochure and a CD containing educational videos pertaining to Pranic healing. Martha Rogers' Science of Unitary Human Beings, the concept of "Nursing as Facilitation of Healing" is central to understanding the role of nurses in promoting health and well-being. In this study, we will use Roger's concept of "nursing as a facilitator of healing" from Pranic Healing method as a facilitator of the healing process. The Pranic advanced protocol will be applied as conceptualized by Master Choa Kok Sui (Sui CK, 2004). Pranic healing protocol applied in this study will be based on the following seven techniques: 1. sensitizing the hands, 2. scanning the Aura, 3. cleansing the aura, 4. increasing the receptivity, 5. energizing with prana, 6. Stabilizing the projected prana and 7. Releasing (Sui choa kok, 2018) (Jois et al., 2018).

For the sampling, after ensuring that children will be ready for sampling, the nurse will be performed venipuncture then, the intervention will be performed in three stages (5 minutes before, during, and 5 minutes after venipuncture ). In the control group, no intervention will be performed, and children only received routine care. Children pain, the arterial oxygen saturation, the number of breaths and pulse rate will be measured and recorded. The venipuncture will be done by a skilled nurse. In order to ensure the consistency of the conditions, the intervention will be scheduled for shifts in which the nurse will be on duty in the ward.

Ethic committee:

The study's aim and methodology will be explained to the participants. Participants will be given the assurance that they can leave the study at any moment without incurring any fees. Finally, the parent and children who voluntarily stated their involvement in the study will provide written informed consent. The study was carried out in accordance with the Declaration of Helsinki's principles (Declaration H, 1964). Moreover, 1. After gaining consent (the experimental and control groups' signed written consent), the participants were informed of the research's goals and placed into groups as project samples. 2. The project units received guarantees that the data is private and won't have any unfavourable effects. 3. It was assured to the project units that doing this yoga has no negative effects. 4. The goals and benefits of the initiative were presented to the authorities, who will also have access to the results upon request. 5. If they agreed, the control group received super brain yoga training. Every participant gave written agreement as a volunteer and acknowledged that they were free to leave the study at any moment. The written consents to participate in the project were received.

Statistical analysis:

The data is entered into spss26 software. Descriptive statistics are performed for quantitative changes with size and quality deviation, and for qualitative changes with frequency and percentage. Chi-square test or Fisher's exact test is used in inferential statistics for several qualities. For quantitative changes, after checking the hypothesis of normality with the Kolmogorov Smirnov test, independent t-tests and repeated measures analysis of variance (ANOVA) or their non-parametric equivalent Mann-Whitney and Wilcoxon tests will be used. A significance level of less than 0.05 is considered for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years experiencing pain during venipuncture
* Willingness of the child and family to cooperate and participate in the research
* No specific mental disorder as reported by the parents
* Not having taken acetaminophen or any other painkillers the night before

Exclusion Criteria:

* Severe restlessness of the child
* Lack of consent from the mother to continue participating in the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Levels During Venipuncture | Pain levels will be measured at three time points: 5 minutes before venipuncture, during venipuncture, and 5 minutes after venipuncture.
  The primary outcome measure will assess changes in pain levels experienced by children during venipuncture. Pain will be evaluated using the Wong-Baker FACES Pain Rating Scale, which is a validated tool for measuring pain in pediatric patients. The Wong-Baker FACES Pain Rating Scale ranges from 0 to 10, with 0 indicating "no pain" and 10 indicating "the worst pain possible." Higher scores represent worse pain outcomes.

SECONDARY OUTCOMES:
Changes in Arterial Oxygen Saturation | Arterial oxygen saturation will be recorded at 5 minutes before venipuncture, during venipuncture, and 5 minutes after venipuncture.
  This secondary outcome measure will evaluate the changes in arterial oxygen saturation levels before, during, and after venipuncture. Oxygen saturation will be monitored using a pulse oximeter.
Changes in Respiratory Rate | Respiratory rate will be measured 5 minutes before venipuncture, during venipuncture, and 5 minutes after venipuncture.
  The respiratory rate of children will be monitored to observe any changes due to the Pranic Healing intervention. The rate will be measured in breaths per minute.
Changes in Pulse Rate | Pulse rate will be recorded at 5 minutes before venipuncture, during venipuncture, and 5 minutes after venipuncture.
  The pulse rate of children will be assessed to detect any variations due to the Pranic Healing intervention. Pulse rate will be measured in beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Pouran Varvani Farahani, PhD, Principal Investigator — PhD student in Pediatric Nursing, Near East University, Faculty of Nursing
Locations (1):
- Near East University, Nicosia, KKTC (Turkish Republic of Northern Cyprus), Cyprus

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Bahrami P, Sheikhan E, Soulari ZS, Golchin M. The Effect of Gentle Touch on Cardiorespiratory Indices and Pain Behaviors Related to Venipuncture and Blood Sampling in Preterm Infants Under Intensive Care. Iran J Nurs Midwifery Res. 2023 Jun 21;28(3):273-279. doi: 10.4103/ijnmr.ijnmr_306_21. eCollection 2023 May-Jun. PMID 37575506
- [Background] Nittur A, Pavan B, Ganapathy R, Dorai VK, Singhal S. Pranic Healing as a Complementary Therapy in Diabetic Foot Ulcer Management: A Randomised, Controlled, Double-Blind Trial. Glob Adv Integr Med Health. 2023 Oct 23;12:27536130231183429. doi: 10.1177/27536130231183429. eCollection 2023 Jan-Dec. PMID 37881236
- [Background] Yilmaz Kurt F, Aytekin Ozdemir A, Atay S. The Effects of Two Methods on Venipuncture Pain in Children: Procedural Restraint and Cognitive-Behavioral Intervention Package. Pain Manag Nurs. 2020 Dec;21(6):594-600. doi: 10.1016/j.pmn.2019.09.002. Epub 2019 Oct 15. PMID 31628067
- [Background] Matourypour P, Zare Z, Mehrzad V, Musarezaie A, Dehghan M, Vanaki Z. An investigation of the effects of therapeutic touch plan on acute chemotherapy-induced nausea in women with breast cancer in Isfahan, Iran, 2012-2013. J Educ Health Promot. 2015 Aug 6;4:61. doi: 10.4103/2277-9531.162380. eCollection 2015. PMID 26430688
- [Background] Alp FY, Yucel SC. The Effect of Therapeutic Touch on the Comfort and Anxiety of Nursing Home Residents. J Relig Health. 2021 Jun;60(3):2037-2050. doi: 10.1007/s10943-020-01025-4. PMID 32415423
- [Background] Gantt M, Orina JAT. Educate, Try, and Share: A Feasibility Study to Assess the Acceptance and Use of Reiki as an Adjunct Therapy for Chronic Pain in Military Health Care Facilities. Mil Med. 2020 Mar 2;185(3-4):394-400. doi: 10.1093/milmed/usz271. PMID 31642490
- See also: Official site for Pranic Healing with information about techniques and training. — http://www.pranichealing.com
- See also: Website for Near East University Faculty of Nursing, providing details about the institution and its research activities. — https://neu.edu.tr/?lang=en
- Available data/document: Study Protocol: NEU-2024-Protocol — https://neu.edu.tr/research/scientific-research-ethics-board/?lang=en — The study protocol will be available through the Near East University research portal. For access, please contact the central research office at Near East University